CLINICAL TRIAL: NCT01015352
Title: A Phase II Study of Azacitidine (Vidaza®) Combined to Epoetin Beta (NeoRecormon®) in IPSS Low-risk and Intermediate-1 MDS Patients, Resistant to ESA
Brief Title: Azacitidine Combined to Epoetin Beta in International Prognostic Scoring System (IPSS) Low-risk and Intermediate-1 Myelodysplastic Syndrome (MDS) Patients, Resistant to Erythropoetin-stimulating Agents (ESA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Celgene Corporation (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-Aza-Epo-2008-01
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2009-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Azacitidine 75mg/sqm SQ per day for 5 days every 28 days for 6 courses and 12 additional maintenance courses in responders.
  Interventions: Drug: Azacitidine
- Arm B (Active Comparator): Azacitidine: 75mg/sqm SQ per day for 5 days every 28 days for 6 courses AND
  Epoetin beta : 60000U weekly SQ injections (to be adapted according to Hb as described above)
  12 additional maintenance courses are planned in responders
  Interventions: Drug: Azacitidine; Drug: Epoetin beta

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 75mg/sqm SQ per day for 5 days every 28 days
  Other Names: Vidaza®
Drug: Epoetin beta — Epoetin beta : 60000U weekly SQ injections
  NeoRecormon®
  Other Names: Epoetin beta : 60000U weekly SQ injections
  Arms: Arm B

SUMMARY:
The study is aimed to treat low-risk MDS patients,who are dependent on red-blood cell transfusion due to disease-related anemia, and who have a proven resistance towards treatment with erythropoetin-stimulating agents (ESA). The study randomizes patients to receive a treatment with the demethylating agent 5-azacytidine alone or in combination with an ESA. The study thus evaluates, if efficacy of 5-azacytidine, notably on the red-blood cell transfusion-dependence is comparable/inferior to a combination treatment with azacitidine and an ESA (that is if 5-azacytidine can overcome the resistance towards ESA). Being a phase II study, the study assesses, duration of erythroid response, overall survival and time to progression as well as toxicity.

DETAILED DESCRIPTION:
Phase II Study of Azacitidine (Vidaza®) Combined to Epoetin Beta (NeoRecormon®) in IPSS Low-risk and Intermediate-1 MDS Patients, Resistant to ESA

The Primary Endpoint of this study is to determine the major erythroid response rate after 6 courses, assessed according to IWG 2000 criteria.

The Secondary Endpoints are to determine the percentage of major HI-E and minor HI-E after 4 and 6 courses according to IWG 2000, the HI-E IWG 2006 criteria, the duration of erythroid response, the red blood cell transfusion independence at 4 and 6 months, the overall survival and time to IPSS progression and the toxicity (NCI-CTAE).

The trial will enroll 98 patients (49 patients per arm)

Treatment in arm A:

Azacitidine 75mg/sqm SQ per day for 5 days every 28 days for 6 courses Dosing of each subsequent course will be adapted according to extrahematological toxicity and cytopenias.

In responders after 6 courses of azacitidine according to IWG 2000 criteria (both minor and major erythroid responses of HI-E) 12 identical additional maintenance courses will be delivered every 28 days, unless relapse occurs (according to IWG 2000 criteria).

Treatment in arm B:

• Azacitidine 75mg/sqm SQ per day for 5 days every 28 days for 6 courses.

(dosing of each subsequent course will be adapted according to extra hematological toxicity and cytopenias) AND

• Epoetin beta : 60000U weekly SQ injections Dosing of epoetin beta will be adapted according to current ASH-ASCO guidelines and black box warning of epoetin beta. Epoetin beta therapy may therefore be interrupted, in case of response to azacitidine, as soon as a hemoglobin level of 12g/dl is achieved on two sequential bimonthly blood count measurements.

A 40% dose reduction of epoetin beta will be required if:

* Hb level rise of 1 g/dl is observed within two weeks
* Hb level exceeds 11g/dl

In responders after 6 courses of azacitidine + epoetin beta, according to IWG 2000 criteria (both minor and major erythroid responses of HI-E) 12 identical additional maintenance courses of azacitidine will be delivered every 28 days, unless relapse occurs (according to IWG 2000 criteria) Epoetin beta will be administered as described above.

In both arms, each subsequent course will be delivered

* In absence of persistent grade >2 non-hematological toxicity
* In absence of rehospitalisation for severe bleeding, infection or febrile neutropenia and non-hematological toxicity following the previous course
* If neutrophil counts are > 1G/l or > 50% of baseline neutrophil counts
* If platelets are > 75G/l or > 50% of baseline platelets counts

In case of persistent cytopenia, blood counts will be at least checked every 2 weeks, and the next course delayed until resolution of cytopenia, as defined above.

In case of persistence of cytopenia beyond day 56 of the preceding course, an new evaluation of the disease, using clinical examination, blood and bone marrow examinations +/- cytogenetics will be mandatory before eventually pursuing azacitidine at lower dosing levels.

ELIGIBILITY:
Inclusion Criteria:

MDS defined as

* RCMD, RA with or without ring sideroblasts
* RAEB 1, or CMML 1, if WBC < 13 G /l according to the WHO classification
* with a low or int-1 IPSS score AND
* primary or secondary resistance to epoetin alpha/ beta (> 60000 U/w) or darbepoetin (> 250ug/w), administered for at least 12 weeks
* requirement of RBC transfusions > 4 U in the previous 8 weeks
* Aged 18 years or more
* Adequate contraception, if relevant
* Negative pregnancy test if relevant
* Written Informed consent
* Ability to participate to a clinical trial and adhere to study procedures
* Health insurance

Exclusion Criteria:

* Therapy-related MDS (after chemo- or radiotherapy for a previous neoplasm or immune disorder)
* Patients with a planned allogeneic bone marrow transplantation
* Creatininemia >1.5 upper normal value or estimated Ccr less than 30ml/mn
* ALAT and ASAT >2.5 upper normal value
* Bilirubin >2N, except unconjugated hyperbilirubinemia due to MDS-related dyserythropoiesis
* Heart failure NYHA > II
* Known allergy to mannitol
* Other tumor, unstable for the last three years, except in situ uterine carcinoma or basal skin tumor
* ECOG > 2
* Life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine the major erythroid response rate after 6 courses, assessed according to IWG 2000 criteria | after 6 courses of treatment in the respective treatment arm

SECONDARY OUTCOMES:
Degree and duration of erythroid response (including red blood cell transfusion independence),overall survival and time to progression and toxicity | after 4 and 6 months of treatment until the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Simone Boehrer, MD, Principal Investigator — Groupe Francophone des Myélodysplasies; Claude Gardin, MD, Principal Investigator — Groupe Francophone des Myélodysplasies
Locations (29):
- France (29):
  - CHU d'Amiens, Amiens
  - Hôpital Angers, Angers
  - Hôpital Avignon, Avignon
  - Hôpital de la Côte Basque, Bayonne
  - Hopital Avicenne, Bobigny
  - Hôpital Boulogne Sur Mer, Boulogne-sur-Mer
  - Hopital Clémenceau, Caen
  - Hôpital le Bocage, Dijon
  - Hôpital Versailles, Le Chesnay
  - Hôpital kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Saint Vincent, Lille
  - Hôpital Huriez, Lille
  - Hôpital Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Paoli-Calmettes, Marseille
  - Hôpital Brabois, Nancy
  - Hôpital Hôtel Dieu, Nantes
  - Hôpital Archet1, Nice
  - Hôpital La Source, Orléans
  - Hôpital Lariboisière, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Maréchal Joffre, Perpignan
  - Hôpital Jean-Bernard, Poitiers
  - Hôpital Reims, Reims
  - Hôpital Henri Becquerel, Rouen
  - Hôpital Hautepierre, Strasbourg
  - Hôpital Purpan, Toulouse

REFERENCES:
- [Derived] Thepot S, Ben Abdelali R, Chevret S, Renneville A, Beyne-Rauzy O, Prebet T, Park S, Stamatoullas A, Guerci-Bresler A, Cheze S, Tertian G, Choufi B, Legros L, Bastie JN, Delaunay J, Chaury MP, Sanhes L, Wattel E, Dreyfus F, Vey N, Chermat F, Preudhomme C, Fenaux P, Gardin C; Groupe Francophone des Myelodysplasies (GFM). A randomized phase II trial of azacitidine +/- epoetin-beta in lower-risk myelodysplastic syndromes resistant to erythropoietic stimulating agents. Haematologica. 2016 Aug;101(8):918-25. doi: 10.3324/haematol.2015.140988. Epub 2016 May 26. PMID 27229713
- See also: (Website of the french group of MDS) — http://www.gfmgroup.org